CLINICAL TRIAL: NCT00160407
Title: Orlistat (Xenical) in the Treatment of Overweight Patients With Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12458; XEN185
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Fatty Liver; Hepatitis
Keywords: nonalcoholic steatohepatitis; enzyme inhibitors; lipase; obesity; insulin resistance
MeSH Terms: conditions — Fatty Liver; Hepatitis; Non-alcoholic Fatty Liver Disease; Obesity; Insulin Resistance | interventions — Orlistat; Diet; CD36 Antigens

INTERVENTIONS:
Drug: Orlistat (Xenical)
Behavioral: 1400 kcal diet (30% fat)

SUMMARY:
The purpose of this study is to determine if orlistat (Xenical) therapy in overweight patients with NASH leads to enhanced weight loss over time, with subsequent improvement in the underlying necroinflammatory and fibrotic changes that are typical of NASH.

DETAILED DESCRIPTION:
Previous studies have suggested that steady weight loss over time will result in improvement in aminotransferases, and more importantly, underlying histopathology in patients with NASH. A total of 50 biopsy-proven NASH patients will be enrolled in a prospective, randomized fashion. Twenty-five patients have been enrolled at the primary study site at Saint Louis University. Recruitment of the next 25 patients is taking place at a study subsite at Brooke Army Medical Center in San Antonio, Texas.

This will be an open-label study comparing an established weight loss program (1400-calorie diet with 30% fat) plus daily vitamin E (800 IU) and a daily multivitamin to the same weight loss program, daily vitamin E (800 IU) and multivitamin, plus orlistat (120 mg), three times daily for 36 weeks.

Data to be collected from prospective patients includes demographic information, such as age, sex, past medical history, medications, height and weight. Biochemical data to be collected from prospective patients includes liver enzymes, measures of insulin resistance to include, insulin levels, lipid panel, hemoglobin A1C, free fatty acids, complete blood count, coagulation studies, and vitamin E levels. Blood will also be collected and stored for markers of inflammation and fibrosis, such as C reactive protein and TNF-alpha. A liver biopsy will be obtained at the completion of the study for both histopathologic analysis and RNA analysis.

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy obtained no more than 24 months before randomization with a pathology report confirming that the histological diagnosis is consistent with NASH
* Compensated liver disease with the following laboratory parameters at the entry visit:

  * Hemoglobin values of greater than or equal to 12 gm/dl for females or 13 gm/dl for males
  * WBC count > 3,000/mm3
  * Neutrophil count > 1,500/mm3
  * Platelets > 70,000/mm3
  * Albumin >3.0 g/dl
* Serum creatinine <1.4mg/dl
* Ability to give informed consent
* Alanine aminotransferase (ALT) greater than or equal to 40 U/L
* BMI > or equal to 27 kg/m2
* Patients who receive orlistat must agree to participate in Xenicare, a free dietary counseling program provided by Roche (sponsor)

Exclusion Criteria:

* Any cause for chronic liver disease other than NASH
* Evidence of decompensated liver disease such as a history of or presence of ascites, bleeding varices, or spontaneous encephalopathy
* History of alcohol consumption of greater than 20 grams per day in the past 2 years
* Prior surgical procedures to include gastroplasty, jejunoileal or jejunocolic bypass
* TPN within the past 6 months
* History of prior organ transplantation
* Concurrent enrollment in other experimental treatment protocols
* Use of ursodeoxycholic acid, rosiglitazone, pioglitazone, or metformin within the 6-month period before enrollment
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is weight loss leading to improvement in the global necroinflammatory and fibrosis scores on liver biopsies. A change of one point in the necroinflammatory grade or fibrosis stage will be considered statistically significant.

SECONDARY OUTCOMES:
BMI,ALT,Serum free fatty acids,HOMA-IR (fasting insulin x fasting glucose/22.4)

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Tetri, MD, Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - Saint Louis University, St Louis, Missouri
  - Brooke Army Medical Center, San Antonio, Texas

REFERENCES:
- [Derived] Harrison SA, Fecht W, Brunt EM, Neuschwander-Tetri BA. Orlistat for overweight subjects with nonalcoholic steatohepatitis: A randomized, prospective trial. Hepatology. 2009 Jan;49(1):80-6. doi: 10.1002/hep.22575. PMID 19053049